CLINICAL TRIAL: NCT03033680
Title: Establishing 18F-PBR06 PET Imaging as a Viable Pharmacodynamic Endpoint in MSA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vikram Khurana, Assistant Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P002373
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: MSA

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple System Atrophy (MSA) (Experimental): Eight subjects with a probable MSA diagnosis will be recruited for this study. Each subject will undergo a [F-18]PBR06 PET scan at baseline, and at 9 months follow-up.
  Interventions: Drug: [F-18]PBR06

INTERVENTIONS:
Drug: [F-18]PBR06 — PET radiopharmaceutical
  Other Names: [18-F]PBR06

SUMMARY:
The specific aims of the study are:

Primary: To determine the presence and regional distribution of microglial activation, as assessed by [F-18]PBR06 PET, in subjects with MSA as compared to healthy controls, at baseline and at 9 months follow-up.

Secondary:

To assess the relationship between microglial activation and clinical progression at baseline and follow-up.

Hypothesis: The working hypothesis is that there is microglial activation in Multiple System Atrophy and that the presence and regional distribution of microglial activation is different in MSA versus healthy controls and correlates with disease severity and comorbidities.

DETAILED DESCRIPTION:
Sixteen subjects with a probable MSA diagnosis will be recruited for this study. A probable MSA diagnosis will be based on the following criteria:

* Autonomic failure involving urinary incontinence (inability to control the release of urine form the bladder, with erectile dysfunction in males) or an orthostatic decrease of blood pressure within 3 min of standing by at least 30 mmHg systolic or 15 mm Hg diastolic and
* Poorly levodopa-responsive Parkinsonism (bradykinesia with rigidity, tremor, or postural instability) or
* A cerebellar syndrome (gait ataxia with cerebellar dysarthria, limb ataxia, or cerebellar oculomotor dysfunction)

Summary:

Subjects will be recruited during routine clinical appointments by their physician or one of the other co-investigators listed on the protocol at the Movement Disorders Clinic, 60 Fenwood Road, Boston, MA. Once the subject gives the informed consent, investigators will be administering standardized questionnaires for assessment of disease severity, comorbidities and/or presence of symptoms, as applicable to a given cohort. In addition, a blood sample will be drawn for genotype testing to identify high affinity, medium affinity, and low affinity binders. Any subjects identified as low affinity binders will be excluded from the study.

Subjects will undergo two PET scans with [F-18]PBR06 at BWH PET scanning facility at 75 Francis Street, Boston, MA. For PET scanning, an intravenous (IV) catheter will be inserted for injection of tracer. In addition, prior to the tracer injection, a second IV catheter may be inserted into the other arm or hand vein on the contralateral side for blood sampling. To increase the usefulness of blood sampling for radiotracer analysis, the hand or arm used for blood sampling may be wrapped in an electrical warmer with the thermostat set at 44°C for approximately 5-10 minutes.The whole PET session will last approximately 120 min. At the time of imaging, the subjects will be positioned in the gantry of a PET camera. A head support will be used to minimize head motion.

Side Effects Monitoring:

No side effects from the radiopharmaceutical are expected. The dose of radiopharmaceutical being administered in this study is below that at which investigators would expect any effect, including physical dependence and addiction. There will be a follow up phone call within 24-72 hours after the PET scans, and again 2 weeks after the PET scans to ensure the subject has not suffered from any side effects. Subjects will be exposed to a small amount of radiation. The radiotracer will be prepared in such a way as to ensure that it is sterile and pyrogen free, and its radiochemical purity (RCP) will be determined using Silica Gel-Instant Thin Layer Chromatography and/or high pressure liquid chromatography (HPLC). In addition, because [F-18]PBR06 is a non-FDA approved radioligand, it's use for this study will be reviewed by Radioactive Drugs Research Committee.

Subject Safety:

Subject monitoring during PET scans will be performed using a 2-way intercom system between the scanner operator and subject and by visual monitoring of the subject through the window into the scan room (the subject is visible to the operator at all times).

Subjects will need to lie still in the PET camera for period of 120 min, and subjects may find it uncomfortable to remain still over this time. Therefore, as mentioned above, subjects will be given the opportunity to take a break for up to 15 minutes after 45 minutes of PET scanning, following which the last 60 minutes of scanning will be completed. A standard head-support device will be used to make the subjects comfortable during the scanning.

If subjects find an intravenous catheter or duration of scanning too uncomfortable, they are free to withdraw from the study at any time.

Recruitment Procedures:

Physicians at Movement Disorders clinic may present the study to a subject during a regular scheduled clinic visit. If the subject is interested in the study, a copy of the consent form will be given. Established Movement Disorders clinic patients may be sent a recruitment letter describing the study and a copy of the consent document. Interested subjects are directed to contact research staff via a telephone number provided in the letter for participation in the study. At the time of the subject's initial screening visit, a licensed physician investigator will answer any questions the subject may have regarding the study and subsequently obtain informed consent. In accordance with NIH guidelines, efforts will be made to attain a mix of study participants, in terms of gender and racial/ethnic representation.

Consent Procedures:

Informed consent will be obtained from the subjects by a licensed physician investigator on the study protocol. Existing Movement Disorders clinic subjects may be sent a letter describing the study and a copy of the consent document. Patients of the clinic may be introduced to the study through fliers posted throughout the clinic. For the PI's own patients, the recruitment letter will be sent several weeks before inquiring about their interest in the study and/or a clinic nurse or a colleague listed on the IRB will introduce the study using the IRB-approved flier in order to avoid the potential for coercion. Interested subjects are directed to contact research staff via a telephone number provided in the letter and on the fliers inviting participation in the study to set up a screening visit. They will have the opportunity to discuss the study with research study staff prior to giving consent as outlined above. Subjects approached for participation in the study during a routine clinical visit will have the opportunity to participate in the study at that time or they may choose to return for participation at another time in the future. All subjects will be informed that they are free to withdraw consent from the study at any time without affecting the quality or type of care that they receive at BWH. Subjects will be informed that they may not qualify for the study if their genetic analysis reveals that they are low affinity binders for TSPO.

Monitoring and Quality Assurance:

During the study period, subjects will be followed by their clinical neurologists for adverse events and disease progression. If problems are reported to their physicians, they will receive care as is normally performed. In addition, the PI will review all laboratory results of tests undergone by the subjects during the study period and help co-ordinate any necessary care with patient's primary providers.

ELIGIBILITY:
Inclusion Criteria:

1. Probable MSA clinical diagnosis.
2. Male and female subjects age 18 to 70 years.
3. Motor symptom onset <2 years prior.
4. Available brain MRI.

Exclusion Criteria:

1. Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
2. Individuals with bipolar disease and schizophrenia
3. Concurrent medical conditions that contraindicate study procedures.
4. Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
5. Claustrophobia
6. Corticosteroid treatment in the past four weeks
7. Non-MRI compatible implanted devices
8. Low Affinity binders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Tissue Volume of Distribution | 1 month
  PET imaging measurement

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Khuana, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Movement Disorders Clinic, 60 Fenwood Road, Boston, Massachusetts, United States